CLINICAL TRIAL: NCT04554433
Title: Disinfection of SARS-COV-2 ( COVID-19 ) in Human Respiratory Tract by Controlled Ethanol Vapor Inhalation Combined With Oral Asprin .
Brief Title: New Treatment for COVID-19 Using Ethanol Vapor Inhalation .
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ragab, Resident of anesthesia and surgical ICU, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20.08.79
Record Dates: First submitted 2020-09-17; First posted 2020-09-18 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Covid-19; Drug Effect
Keywords: COVID-19; Clinical trial; Ethyl alcohol vapor inhalation
MeSH Terms: conditions — COVID-19 | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: * (A) group: will receive the new protocol .
  * (B) group: Will receive the standard protocol .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): A ) Treatment group will receive a combination of Asprin in anti - inflammatory dose and controlled ethanol vapor inhalation in concentraions and technique according to their medical condition .
  Interventions: Drug: Ethanol with Asprin
- Control (No Intervention): B ) Control group : will receive the standard protocol . Data collection will include : sociodemographic data , clinical history , results of follow up ( daily or according to clinical situation ) Follow up : to record any side effects of drugs , and swab will be taken for PCR .

INTERVENTIONS:
Drug: Ethanol with Asprin — Group ( A ) which will receive the new protocol will be categorized into sub-groups according to the medical conditions , inclusion criteria , investigations and symptoms .
  1. Inhaling alcohol vapor through nostrils .
  2. Inhalation of Alcohol vapor driven by Oxygen .
  3. Inhalation of Alcohol vapor driven by oxygen in case of ARDS.
  4. Ethyl Alcohol infusion into the airway . Investigations will be made before starting the protocol and follow up data will be collected every day .
  Follow up test will be done according to the schedule . PCR test will be done according to the duration of each technique to evaluate the final results .
  Other Names: Controlled ethanol vapor inhalation combined with oral Asprin .
  Arms: Intervention

SUMMARY:
Since ARDS is a major complication of COVID - 19 with subsequent formation of non-cardiogenic pulmonary edema , worsening the oxygenation of the patients and foamy and even bloody sputum formation, so the idea is to use alcohol inhalation as it reduce surface tension on the alveoli and markedly decrease sputum formation with improvement on oxygenation beside its cytolethal effect on virus lipid bilayer.

A lot of researches and publications proved the role of alcohol inhalation in treatment of pulmonary edema. Alcohol inhalation may has inflammatory effect and dangerous effect on patients but this can be controlled by the actual concentration used and the way we use it according to general condition of the patient and with the help of anti - inflammatory action of Asprin .

DETAILED DESCRIPTION:
Corona viruses can cause diseases in both animals and humans. Many of them typically infect upper respiratory tract with minor symptoms. However, three corona viruses can infect lower respiratory tract and cause fatal pneumonia; which are severe acute respiratory syndrome corona virus (SARS-CoV), Middle East respiratory syndrome coronavirus (MERS-CoV) and ( SARS-CoV-2). SARS-CoV-2 shares 78% similarity of genetic material with SARS-CoV.

Pathophysiology of both viruses are closely similar, with destructive inflammatory response resulting in airway damage. That's why, disease severity in patients depends, not only on the viral infection, but also on the host response.

In many cases, this will resolve the infection. However, in other cases, immune response dysfunctions and causes severe lung and systemic pathology ending to ARDS and respiratory failure .

Treatment according to this protocol will be focused on using Asprin to decrease inflammatory reaction weather from the virus or after using alcohol.

Alcohol will be used by different methods and concentration in order to decrease surface tension on alveoli , decreasing foamy sputum secretion , increasing vascular permeability and improving oxygenation .

Also the investigator will use it as a prophylaxis for health care workers to disinfect the virus as soon as possible while it is present in nasal mucosa and upper airway.

Patients will be classified according to inclusion and exclusion criteria and will be divided into groups and they will receive the protocol as it is designed in concentrations and techniques suitable for their medical condition .

In this trial , The investigator will use 4 method to administrate Ethyl Alcohol to the patient by different concentrations .

1. Inhaling alcohol vapor through nostrils .
2. Inhalation of Alcohol vapor driven by Oxygen .
3. Inhalation of Alcohol vapor driven by oxygen in case of ARDS.
4. Ethyl Alcohol infusion into the airway . In each method , the patient will be prepared for one day before starting the protocol by prophylactic antibiotic , anti - inflammatory , mucolytic and bronchodilators .

Investigations will be made before starting for follow up of the results .

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 - 60
* Confirmed COVID-19 positive with PCR test .
* Admitted to Mansoura university quarantine hospital ..
* Fever ≥ 38
* Respiratory rate ≥ 20
* Myalgia , Arthralgia and Sore throat .
* Radiological findings consisting with COVID-19 .
* Welling to participate and able to give fully informed consent. Specific inclusion criteria according to the concentration and method :-

  * Inhalation of Alcohol vapor driven by Oxygen Respiratory distress ( Dyspnea - Orthopnea ) Spo2 : 65 - 85 ABG : Respiratory Alkalosis due to dyspnea and tachypnea PaO2 / FIO2 ratio > 300 mmHg under the condition in the hospital room (Moderate illness).
  * Inhalation of Alcohol vapor driven by oxygen in case of ARDS. Respiratory failure . CT : lobar collapse and nodules Non cardiogenic pulmonary edema excluded by ECHO or signs of overload . PaO2 / FIO2 ratio 101 - 300 mmHg on CPAP or Vent . ( Mild to moderate ARDS)
  * Ethyl Alcohol infusion into the airway PaO2 / FIO2 ratio ≤ 100 mmHg ( Sever ARDS )

Exclusion Criteria:

* Absence of any item from inclusion criteria
* Pregnancy .
* Signs of dehydration , Sepsis or shortness of breathing.
* Asthmatic patients .
* COPD .
* Smokers ≥ 10 years .
* Hypersensitivity to Alcohol

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Disinfection of COVID-19 in human respiratory tract . | Negative PCR test within 7 days from starting the protocol .
  Destruction of COVID-19 in human respiratory tract and treatment of the patients with COVID 19 and Negative PCR test .

SECONDARY OUTCOMES:
Improvement of general condition of mechanically ventilated patients confirmed COVID-19 positive .. | Negative PCR test within 10 days from starting the protocol .
  Decrease mortality rate of mechanically ventilated patients with COVID-19 . Protection of health care workers . Negative PCR test .